CLINICAL TRIAL: NCT01136759
Title: Expanded Safety Investigation of Tenofovir 1% Gel in Pregnancy and Lactation
Brief Title: Tenofovir Gel in Pregnancy and Lactation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MTN-008; 10805 (Registry Identifier: DAIDS Protocol #); MTN 008; 5U01AI068633-04 (NIH)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2014-09

CONDITIONS: HIV Infections
Keywords: Prevention; Microbicide; Mother-to-Child-Transmission; Pregnancy
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pregnancy cohort, placebo (Placebo Comparator): Pregnant women will receive placebo gel.
  Interventions: Other: Placebo gel
- Lactation cohort, tenofovir gel (Experimental): Lactating mothers will receive tenofovir gel.
  Interventions: Drug: Tenofovir 1% gel
- Pregnancy cohort, tenofovir gel (Experimental): Pregnant women will receive tenofovir gel.
  Interventions: Drug: Tenofovir 1% gel

INTERVENTIONS:
Drug: Tenofovir 1% gel — One applicator of tenofovir 1% gel administered vaginally for 7 consecutive days
  Other Names: Tenovofir disproxil fumate; TDF
  Arms: Lactation cohort, tenofovir gel; Pregnancy cohort, tenofovir gel
Other: Placebo gel — One applicator of placebo gel administered vaginally for 7 consecutive days
  Arms: Pregnancy cohort, placebo

SUMMARY:
Tenofovir 1% gel is an investigational vaginal microbicide intended to reduce the risk of transmission of HIV. Pregnant women and mothers who have recently given birth often maintain sexual activity, and research has shown that they may be at greater risk of HIV infection during pregnancy. Microbicides may be able to prevent HIV infection during pregnancy, which would also prevent fetal exposure to HIV. This study will test the safety of using tenofovir 1% gel in healthy, pregnant women and healthy, breastfeeding women.

DETAILED DESCRIPTION:
Microbicides are substances, like gels or foams, being developed that can be applied before intercourse to prevent transmission of HIV. Research has shown that pregnant women are still at risk of sexual transmission of HIV, and some research has suggested that pregnant women may be at increased risk of HIV infection. Microbicides may also aid in preventing mother-to-child transmission of HIV, because they might be a feasible alternative to oral or intravenous medications in regions where these methods are difficult to implement. In tests on healthy women the vaginal microbicide tenofovir 1% gel has been safe and well tolerated. This study will test the safety of tenofovir 1% gel in healthy, pregnant women and healthy, lactating women.

Participation in this study will last approximately 3 to 10 weeks. Pregnant women will be followed until approximately 2 weeks after delivery of their children, and lactating women will be followed for 3 weeks. Pregnant women will be given either the tenofovir 1% gel or a placebo gel to be applied daily for 7 days. Groups of pregnant women will be further divided according to how late into pregnancy they enroll.

Pregnant women will have study visits at enrollment, 6 days after enrollment, and at delivery. They will also participate in phone assessments 1, 3, and 14 days after enrollment and at delivery.

Lactating women will be given tenofovir 1% gel and have study visits at enrollment and 6 days after enrollment. They will also participate in phone assessments 1, 3, and 14 days after enrollment.

All participants will complete blood tests, physical exams, and assessments of adverse events.

ELIGIBILITY:
Pregnancy cohort, inclusion criteria:

* Willing and able to provide written informed consent to be screened for and take part in the study, including participation of the infant after delivery
* Willing and able to provide adequate locator information
* Willing and able to communicate in written and spoken English
* HIV uninfected
* Current pregnancy that is viable and a singleton
* Gestational age consistent with the following guidelines:

  * For Pregnancy Cohort Group 1, between 37 0/7 and 39 1/7 weeks (inclusive) at the enrollment visit (Day 0)
  * For Pregnancy Cohort Group 2, between 34 0/7 and 36 6/7 weeks (inclusive) at the enrollment visit (Day 0)
* Pap result consistent with Grade 0 or satisfactory evaluation of a non-Grade 0 Pap result, per clinical judgment of site investigator or record (IoR)/designee), in the 12 calendar months prior to enrollment
* Willing to abstain from using nonprescribed intravaginal products and practices (including douching and sex toys) or other investigational agent or device during study participation

Pregnancy cohort, exclusion criteria:

* History of adverse reaction to any component of tenofovir 1% gel
* Enrollment in any other investigational drug or device trial within 30 days prior to the enrollment visit (Day 0)
* Currently breastfeeding
* Use of vaginal medications within 48 hours prior to screening or enrollment (Day 0) (participant may return to complete study procedures after 48 hours have passed since use of vaginal medication)
* Documented to have any of the following during the current pregnancy:

  * Ultrasound evidence of significant fetal congenital anomaly (in the opinion of the IoR or designee)
  * Known rupture of the amniotic membranes
  * Known placental/fetal abnormalities that could affect placental transfer (e.g., placental abruption, placenta previa, placenta accreta, intrauterine growth restriction, two-vessel cord, etc.)
  * Known maternal disease with predictable negative effect on placental function (e.g., hypertension, diabetes mellitus, collagen vascular disease)
* Laboratory abnormalities noted at screening, as specified in study protocol
* Diagnosis of sexually transmitted infection (STI), including chlamydia, gonorrhea, and/or trichomoniasis, in the past 8 weeks prior to enrollment (Day 0), as assessed by participant report or review of medical record
* Symptomatic vaginitis, including bacterial vaginosis (BV) and vulvovaginal candidiasis (asymptomatic evidence of BV and/or yeast is not exclusionary) at the time of enrollment (Day 0)
* Clinically apparent pelvic exam finding of Grade 2 or higher (observed by study staff) at the enrollment visit
* Use of oral and/or vaginal preparations of antibiotic or antifungal medications at screening or within 7 days of enrollment (Day 0)
* Any social or medical condition that, in the investigator's opinion, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Lactation cohort, inclusion criteria:

* Willing and able to provide written informed consent to be screened for and take part in the study
* Willing and able to provide adequate locator information
* Willing and able to communicate in spoken and written English
* HIV uninfected
* At enrollment, currently primarily breastfeeding a single healthy infant between the ages of 4 and 26 weeks (inclusive)
* Intending to breastfeed during the period of anticipated study participation
* Using an effective method of contraception at enrollment (Day 0) into lactation cohort and intending to use an effective method for the duration of scheduled study participation
* Pap result consistent with Grade 0 or satisfactory evaluation of non-Grade 0 Pap result, per clinical judgment of site IoR/designee, in the 12 calendar months prior to enrollment (Day 0)
* Willing to abstain from using nonprescribed intravaginal products and practices (including douching and sex toys) or other investigational agent or device during study participation

Lactation cohort, mother exclusion criteria:

* Participation in pregnancy cohort
* Infant excluded from participation
* History of adverse reaction to any component of tenofovir 1% gel
* Participation in investigational drug or device trial within 30 days prior to the enrollment visit (Day 0)
* Use of vaginal medication(s) within 48 hours prior to screening or enrollment (Day 0) (participant may return to complete study procedures after 48 hours have passed since use of vaginal medication)
* More than two infant feedings in a single day with nutrition other than own breast milk (e.g., formula, solids) within 7 days prior to screening or enrollment (Day 0)
* At the time of enrollment (Day 0), participant report or clinical evidence of insufficient milk supply or mastitis, according to the judgment of the IoR/designee
* Any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, or immunologic disorder or infectious disease, as determined by the IoR/designee
* Certain laboratory results, as specified by study protocol
* Diagnosis of STI, including chlamydia, gonorrhea, and/or trichomoniasis, in the 8 weeks prior to enrollment (Day 0), as assessed by participant report or review of medical record
* Symptomatic vaginitis, including BV and vulvovaginal candidiasis (asymptomatic evidence of BV and/or yeast is not exclusionary) at the time of enrollment (Day 0)
* Any of the following findings at enrollment:

  * Incomplete postpartum involution of the uterus
  * Clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff)
* Use of oral and/or vaginal preparations of antibiotic or antifungal medications at screening or within 7 days of enrollment (Day 0)
* Any social or medical condition that, in the investigator's opinion, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Lactation cohort, infant inclusion criteria:

* Mother consents for participation of both self and infant in lactation cohort
* In general good health, as determined by clinical judgment of IoR/designee
* Between the ages of 4 and 26 weeks (inclusive) at both screening and enrollment

Lactation cohort, infant exclusion criteria:

* Any social or medical condition that, in the investigator's opinion, would make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 232 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in pregnant women | Measured at 2 weeks post-delivery
  Safety and tolerability in pregnant women are assessed by number of specific Grade 2 or greater adverse events in laboratory abnormalities, genital/pelvic signs/symptoms, or pregnancy complications
Safety and tolerability in infants, defined as no intensive care admission greater than 24 hours and no sepsis | Measured at 2 weeks post-delivery
Safety and tolerability in lactating women, defined as specific Grade 2 or greater adverse events in laboratory abnormalities or genital/pelvic signs/symptoms | Measured at Day 14
  Safety and tolerability in lactating women are assessed by number of specific Grade 2 or greater adverse events in laboratory abnormalities or genital/pelvic signs/symptoms
Safety and tolerability in infants of lactating mothers | Measured at Day 14
  Safety and tolerability in infants of lactating mothers is defined as no inpatient admission (confirmed on review of medical records) with diagnosis of adverse event (AE) judged to be related to study product
Tenofovir levels in maternal blood or breast milk | Measured at Day 6 or delivery, depending on cohort

SECONDARY OUTCOMES:
Presence of tenofovir in blood among infants of participants in the pregnancy and lactation cohorts | Measured at Day 6 or delivery, depending on cohort
Impact of tenofovir gel exposure on the presence of select organisms associated with neonatal sepsis among participants in the pregnancy cohort, (e.g., Group B β-hemolytic streptococcus, Escherichia coli) | Measured at Day 6
Adherence to daily use of tenofovir 1% gel for 7 days and its acceptability among pregnant and lactating women | Measured at Day 6

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Alabama CRS, Birmingham, Alabama
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Rohan LC, Moncla BJ, Kunjara Na Ayudhya RP, Cost M, Huang Y, Gai F, Billitto N, Lynam JD, Pryke K, Graebing P, Hopkins N, Rooney JF, Friend D, Dezzutti CS. In vitro and ex vivo testing of tenofovir shows it is effective as an HIV-1 microbicide. PLoS One. 2010 Feb 19;5(2):e9310. doi: 10.1371/journal.pone.0009310. PMID 20174579
- [Background] Cranage M, Sharpe S, Herrera C, Cope A, Dennis M, Berry N, Ham C, Heeney J, Rezk N, Kashuba A, Anton P, McGowan I, Shattock R. Prevention of SIV rectal transmission and priming of T cell responses in macaques after local pre-exposure application of tenofovir gel. PLoS Med. 2008 Aug 5;5(8):e157; discussion e157. doi: 10.1371/journal.pmed.0050157. PMID 18684007